CLINICAL TRIAL: NCT01619709
Title: Amyloid Imaging and Cognitive Impairment After Intracerebral Hemorrhage
Acronym: COGHIC-AV45
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Collaborators: Avid Radiopharmaceuticals (Industry); Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 11 223 02; AOL 2011 (Other: CHU de Toulouse)
Record Dates: First submitted 2012-06-12; First posted 2012-06-14 (Estimated); Last update posted 2018-09-21 (Actual); Status verified 2018-09

CONDITIONS: Intracerebral Hemorrhage
Keywords: Intracerebral Hemorrhage; Cerebral Amyloid angiopathy; Amyloid imaging; 18F-AV-45
MeSH Terms: conditions — Cerebral Hemorrhage; Cerebral Amyloid Angiopathy | interventions — florbetapir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- lobar hemorrhage group (Other): PET AV-45 in patients with cortical or corticosubcortical hemorrhage (involving predominantly the cortex and underlying white matter)
  Interventions: Other: Pet AV-45
- deep hemorrhage group (Other): PET AV-45patients with subcortical hemorrhage (involving predominately the basal ganglia, periventricular white matter, or internal capsule).
  Interventions: Other: Pet AV-45

INTERVENTIONS:
Other: Pet AV-45 — AV-45 (Florbetapir F 18) : Bolus of 5 MBq/kg IV ; A 10-minutes Pet scan acquisition Starts at 50 minutes after injection.
  Other Names: PET AV-45 (Florbetapir F 18) Cerebral Amyloid imaging

SUMMARY:
To evaluate Pet AV-45 Amyloid imaging in the etiological diagnosis of primary non traumatic intracerebral hemorrhage (Cerebral Amyloid Angiopathy and hypertension related hemorrhage).We hypothesize that patients with lobar hemorrhage (probably related to Cerebral Amyloid Angiopathy) will have a greater AV45 cortical binding than patients with deep hemorrhage (probably related to hypertension).

DETAILED DESCRIPTION:
Cerebral Amyloid Angiopathy (CAA) and hypertension related hemorrhage are the main causes of non traumatic primary intracerebral hemorrhage. In vivo diagnosis of these two cerebral diseases may be difficult and is based on hematoma location and pattern of cerebral microbleeds (CMB) distribution. We aimed to evaluate a multimodal approach including brain MRI, Pet AV-45 Amyloid imaging and neuropsychological assessment to improve etiological diagnosis of primary intracerebral hemorrhage. 70 patients with acute primary non traumatic intracerebral hemorrhage will be prospectively included and two groups will be compared: lobar hemorrhage group and deep hemorrhage group. Brain MRI, Pet AV-45 Cerebral Amyloid imaging (during the first month) and neuropsychological assessment (Three months later) are performed. Differences between the two groups are evaluated for AV45 cortical binding, CMB distribution, White Matter Lesions and cognitive profile.

ELIGIBILITY:
Inclusion Criteria:

* Age : 40-90 years,
* Non traumatic primary intracerebral hemorrhage during acute phase (less than 30 days from hemorrhage onset) confirmed on brain imaging (CT and/or MRI).
* Correct visual, hearing and language functions to perform neuropsychological tests.
* Written consent of patient

Exclusion Criteria:

* Secondary causes of intracerebral hemorrhage : vascular malformations (Arteriovenous malformation, intracranial aneurysm, Cavernous angioma, dural arteriovenous fistula), cerebral venous thrombosis, intracranial neoplasm, coagulopathy, vascularitis, Cocaine or alcohol use, Hemorrhagic ischemic stroke.
* Pregnancy
* Contraindication to MRI
* progressive neoplasm
* Cognitive impairment secondary to progressive neurological disease
* Depression,
* Drug addiction

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2012-01; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Pet-AV45 cortical binding | Acute phase of intracerebral hemorrhage ie during the first month after hemorrhage onset.
  Method of administration: a bolus IV injection (less than 1 minute of injection time) of 5 MBq / kg with a maximum of 370MBq. The activity corresponding to a 70 kg individual is 350 MBq and corresponds to an effective dose of 12.25mSv (0.035mSv/MBq)

SECONDARY OUTCOMES:
cerebral microbleeds number and distribution on T2EG MRI sequence | Acute phase of intracerebral hemorrhage ie during the first month
  Review safe after checking against usual contraindications (pacemaker, ocular foreign body), painless, lasting about 45 minutes, during which a detailed analysis of the brain will be performed
White Matter Lesions Volume on 3D-FLAIR MRI sequence | Acute phase of intracerebral hemorrhage ie during the first month
  Review safe after checking against usual contraindications (pacemaker, ocular foreign body), painless, lasting about 45 minutes, during which a detailed analysis of the brain will be performed
Cortical thickness and hippocampal volume on 3D-T1 MRI sequence | Acute phase of intracerebral hemorrhage ie during the first month
  Review safe after checking against usual contraindications (pacemaker, ocular foreign body), painless, lasting about 45 minutes, during which a detailed analysis of the brain will be performed
Neuropsychological performances | three months after hemorrhage onset.
  a neuropsychological examination (tests of memory, language and attention) will be realized. This examination will last approximately 60 minutes and take place in consultation with neurology

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Raposo, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Service de neurologie, Toulouse, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Planton M, Pariente J, Nemmi F, Albucher JF, Calviere L, Viguier A, Olivot JM, Salabert AS, Payoux P, Peran P, Raposo N. Interhemispheric distribution of amyloid and small vessel disease burden in cerebral amyloid angiopathy-related intracerebral hemorrhage. Eur J Neurol. 2020 Aug;27(8):1664-1671. doi: 10.1111/ene.14301. Epub 2020 May 31. PMID 32394598
- [Derived] Planton M, Saint-Aubert L, Raposo N, Branchu L, Lyoubi A, Bonneville F, Albucher JF, Olivot JM, Peran P, Pariente J. High prevalence of cognitive impairment after intracerebral hemorrhage. PLoS One. 2017 Jun 1;12(6):e0178886. doi: 10.1371/journal.pone.0178886. eCollection 2017. PMID 28570698